CLINICAL TRIAL: NCT05301946
Title: Application of the ICF Core Set for Cognitive Function, Quality of Life and Mobility in Stroke Patients
Brief Title: Application of the ICF Core Set in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Güzin Kara, Research Assistant, Pamukkale University
Other Study IDs: 60116787-020/9175
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Paralysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: The created-ICF Core Set for Stroke including activitiy, participation, and environmental factors was used show the meaningfulness of the clinical outcome measurements. The correlation of the created-ICF Core Set for Stroke's items and the outcome measurements were analyzed through Spearman or Pearson correlation analysis.
  Interventions: Other: Outcome Measurements

INTERVENTIONS:
Other: Outcome Measurements — The 24-item ICF Core Set for Stroke, Standardized Mini-Mental State Examination, Stroke Impact Scale, Rivermead Mobility Index, and Home Safety Checklist were applied to the stroke patients. The assessment period took one hour.

SUMMARY:
Sixty patients with stroke were applied a-24-item ICF Core Set for Stroke, Standardized Mini-Mental State Examination(SMMSE), Stroke Impact Scale Version(SIS), Rivermead Mobility Index(RMI) and Home Safety Checklist(HSCL). Spearman and Pearson correlation analysis was used to show the relation between the items of the scales and the ICF Core Set for Stroke items.

DETAILED DESCRIPTION:
Fourty men and twenty women stroke patients were included in this study.The demographics and clinical information of the participants were recorded. A physiotherapist created an ICF Core Set for Stroke for the study. The ICF Core Set for Stroke was used to show the significant relationship with Standardized Mini-Mental State Examination, Stroke Impact Scale Version 3.0, and Rivermead Mobility Index. The duration of the assessment varied between 1 hour and 1.5 hours depending on the participant.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 25-80,
* Having a single stroke,
* Not having any other condition affecting the evaluation such as aphasia, consciousness disorders, or other neurological diseases.

Exclusion Criteria:

* . Stroke patients who did not complete the evaluations.

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 men, 20 women stroke patients who met the inclusion criteria. were included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Standardized Mini-Mental State Examination | One year
  This scale was used to assess the cognitive status of stroke patients. The maximum score of SMMSE is 30 points.
Stroke Impact Scale | One year
  This scale was used to assess the quality of life in stroke patients. Each domain is scored from 0 to 100.
Rivermead Mobility Index | One year
  This scale was used to assess the mobility levels of stroke patients. The minimum and maximum scores are between 0-15.
Home Safety Checklist | One year
  Ten items of this scale were used to assess the home safety status. The HSCL is scored between 0-65.
A 24-item ICF Core Set for Stroke | One year
  The core set was created and consisted of 24 ICF items. Each category is scored between 0 - 4 and 8, or 9.

CONTACTS AND LOCATIONS:
Overall Officials: Güzin Kara, Ph.D., Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kınıklı/Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tarvonen-Schroder S, Hurme S, Laimi K. The World Health Organization Disability Assessment Schedule (WHODAS 2.0) and the WHO Minimal Generic Set of Domains of Functioning and Health versus Conventional Instruments in subacute stroke. J Rehabil Med. 2019 Oct 4;51(9):675-682. doi: 10.2340/16501977-2583. PMID 31402390
- [Background] Sumathipala K, Radcliffe E, Sadler E, Wolfe CD, McKevitt C. Identifying the long-term needs of stroke survivors using the International Classification of Functioning, Disability and Health. Chronic Illn. 2012 Mar;8(1):31-44. doi: 10.1177/1742395311423848. Epub 2011 Oct 24. PMID 22025770
- [Background] Yarar F, Cavlak U, Basakci Calik B. Applying the International Classification of Functioning, Disability, and Health in children with low vision: differences between raters. Turk J Med Sci. 2016 Dec 20;46(6):1694-1699. doi: 10.3906/sag-1506-152. PMID 28081311